CLINICAL TRIAL: NCT02171260
Title: A Phase 1 Study of Eribulin Mesylate, a Novel Microtubule Targeting Chemotherapeutic Agent in Children With Refractory or Recurrent Solid Tumors (Excluding CNS), Including Lymphomas
Brief Title: This is a Phase 1 Study of Eribulin Mesylate in Pediatric Participants With Recurrent or Refractory Solid Tumors (Excluding [Central Nervous System] CNS), Including Lymphomas
Acronym: BOLD 113
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-113 (ADVL1314)
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-06

CONDITIONS: Pediatrics; Solid Tumors
Keywords: Tumors; Lymphomas; Solid Tumors; Pediatric
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eribulin Mesylate (Experimental): Eribulin mesylate will be administered intravenously on Days 1 and 8 of each 21-day cycle. A cycle of therapy is considered to be 21 days. The starting dose for eribulin mesylate will be at 1.1 milligram per square meter (mg/m^2) (Dose Level 1), which is approximately 80% of the adult MTD, and will be escalated up to no more than 2.2 mg/m^2.
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate will be administered intravenously on Days 1 and 8 of each 21-day cycle.
  Other Names: E7389

SUMMARY:
This is a Phase 1 study of eribulin mesylate in pediatric participants with recurrent or refractory solid tumors (excluding CNS), including lymphomas. Eribulin mesylate will be administered intravenously, once per day on Days 1 and 8 of a 21-day cycle. This study aims to determine the maximum tolerated dose (MTD) and/or the Recommended Phase 2 Dose (RP2D) of this regimen in Part A1 (participants greater than or equal to [>=] 12 months and less than [<] 18 years). Part A2 will enroll infants (greater than [>] 6 months and <12 months) one dose level behind the dose level at which participants in Part A1 are enrolling, in order to maximize safety for infant participants. Additionally, this study aims to describe the toxicities and the pharmacokinetics of eribulin mesylate when administered to children. In a preliminary manner, the antitumor effect of eribulin mesylate will also be described.

ELIGIBILITY:
Inclusion Criteria

* Participants must be >=12 months and <18 years of age at the time of study enrollment (Part A1).
* Participants must be >6 months and <12 months of age at the time of study enrollment (Part A2). Participants will enroll one dose level behind the dose level at which participants in Part A1 are enrolling.
* Participants with refractory or recurrent solid tumors or lymphomas, excluding CNS tumors, are eligible. Participants must have had histologic verification of malignancy at original diagnosis or relapse. Participants with primary CNS tumors, known CNS metastases, or a prior history of CNS metastases are not eligible.
* Participants must have either measurable or evaluable disease.
* Participants current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Karnofsky >= 50% for participants >16 years of age and Lansky >=50 for participants less than or equal to (<=)16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Participants must have fully recovered from the acute toxic effects of all prior anticancer chemotherapy.

  1. Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
  2. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (example Neulasta) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  3. Biologic (anti-neoplastic agent): At least 14 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 14 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  4. Immunotherapy: At least 42 days after the completion of any type of immunotherapy, example tumor vaccines.
  5. Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody.
  6. X-ray telescope (XRT): At least 14 days after local palliative XRT (small port); At least 150 days must have elapsed if prior total body irradiation(TBI), craniospinal and/or entire spinal XRT or if >=50% radiation of pelvis; At least 42 days must have elapsed if other substantial bone marrow (BM) radiation.
  7. Stem Cell Infusion without TBI: No evidence of active graft versus host disease and at least 84 days must have elapsed after transplant or stem cell infusion.
* Adequate Bone Marrow Function Defined as:

  1. Peripheral absolute neutrophil count (ANC) >=1000 per cubic millimeter (/mm^3).
  2. Platelet count >=100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
  3. Hemoglobin (Hb) at least 8 gram per deciliter (g/dL) at baseline (blood transfusions are allowed during the screening period to correct Hb values less than 8 g/dL).

All participants enrolled on the study must be evaluable for hematologic toxicity.

* Adequate Renal Function Defined as:

  1. Creatinine clearance or radioisotope glomerular filtration rate (GFR) >=70 milliliter per minute (ml/min) per (/) 1.73 square meter (m^2) or
  2. A serum creatinine milligram per deciliter (mg/dL) based on age/gender as follows:

     1. 6 months to <1 year: male, 0.5; female, 0.5
     2. 1 to < 2 years: male, 0.6; female, 0.6
     3. 2 to < 6 years: male, 0.8; female, 0.8
     4. 6 to < 10 years: male, 1; female, 1
     5. 10 to < 13 years: male, 1.2; female, 1.2
     6. 13 to < 16 years: male, 1.5; female, 1.4
     7. >=16 years: male, 1.7; female, 1.4

        The threshold creatinine values were derived from the Schwartz formula for estimating GFR (Schwartz et al., 1985) utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC).
* Adequate Liver Function Defined as:

  1. Bilirubin (sum of conjugated + unconjugated) <=1.5 * upper limit of normal (ULN) for age
  2. serum glutamic-pyruvic transaminase (SGPT) (alanine transaminase [ALT]) <=110 units per liter (U/L). For the purpose of this study, the ULN for SGPT is 45 U/L.
  3. Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) <= 125 U/L. For the purpose of this study, the ULN for SGOT is 50 U/L.
  4. Serum albumin >= 2 g/dL
* Adequate Cardiac Function Defined as:

  1. Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study
  2. Corrected QT interval (QTc) <= 480 millisecond (msec) Note: Participants with Grade 1 prolonged QTc (450-480 msec) at the time of study enrollment should have correctable causes of prolonged QTc addressed if possible (that is, electrolytes, medications).
* All participants and/or their participants or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines. Participants must be willing to comply with all aspects of the protocol.
* Participants with known human immunodeficiency virus (HIV) who have CD4+ T cell counts greater than or equal to 500 cells/m^3 and who do not require antiretroviral therapy are eligible.

Exclusion Criteria

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective double barrier contraceptive method for the entire period in which they are receiving protocol therapy and up to 6 months after treatment.
* Concomitant Medications

  * Participants receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible.
  * Participants who are currently receiving another investigational drug are not eligible.
  * Participants who are currently receiving other anticancer agents are not eligible.
  * Participants who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial.
  * Participants who are receiving drugs that prolong the QTc are not eligible.
* Participants who have received prior therapy with eribulin mesylate are not eligible.
* Participants with hypersensitivity to excipients of the study drug are not eligible. The excipients are ethanol, hydrochloric acid, sodium hydroxide and water for injection.
* Participants who have a prior history of viral hepatitis (B or C) as demonstrated by positive serology (presence of antigens) or have an uncontrolled infection requiring treatment are not eligible.
* Participants with greater than Grade 1 peripheral sensory neuropathy or greater than Grade 1 peripheral motor neuropathy graded according to the Modified ("Balis") Pediatric Scale of Peripheral Neuropathies are not eligible.
* Cardiac Pathology

  * Participants with known congestive heart failure, symptomatic or left ventricle (LV) ejection fraction 50% or shortening fraction less than 27% are not eligible.
  * Participants with congenital long QT syndrome, bradyarrhythmias, or QTc greater than 480 msec are not eligible.
* CNS Disease

  * Participants with primary CNS tumors are not eligible.
  * Participants with prior history of or known metastatic CNS disease involvement are not eligible. (Note: CNS imaging for participants without a known history of CNS disease is only required if clinically indicated).
* Participants who have had or are planning to have the following invasive procedures are not eligible:

  * Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to enrollment.
  * Central line placement or subcutaneous port placement is not considered major surgery but must be placed at least 3 days prior to enrollment for external lines (with example, Hickman or Broviac) and at least 7 days prior to enrollment for subcutaneous port.
  * Core biopsy within 7 days prior to enrollment.
  * Fine needle aspirate within 7 days prior to enrollment. NOTE: For purposes of this study, bone marrow aspirate and biopsy are not considered surgical procedures and therefore are permitted within 14 days prior to start of protocol therapy.
* Participants with known bone marrow involvement are not eligible.
* Participants who have received a prior solid organ transplantation are not eligible.
* Participants who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Childrens Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Cancer Center-Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in the United States from 31 July 2014 to 28 January 2016.
Pre-assignment Details: In Part A1, a total of 23 participants of greater than or equal to (>=) 12 months were enrolled, of which 22 were treated in the study. In Part A2, the study was open for the enrolment of infant participants of less than 12 months of age, however no participants were enrolled into this part.
Groups:
- Part A1: Eribulin Mesylate 1.1 mg/m^2: Participants received eribulin mesylate (E7389) 1.1 milligram per square meter (mg/m^2), intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 4 cycles, or until progressive disease (PD) or unacceptable toxicity or drug related dose-limiting toxicities (DLT's).
- Part A1: Eribulin Mesylate 1.4 mg/m^2: Participants received eribulin mesylate 1.4 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 8 cycles, or until PD or unacceptable toxicity or drug related DLT's.
- Part A1: Eribulin Mesylate 1.8 mg/m^2: Participants received eribulin mesylate 1.8 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 5 cycles, or until PD or unacceptable toxicity or drug related DLT's.
- Part A1: Eribulin Mesylate PK Expansion: Participants received eribulin mesylate 1.4 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 2 cycles, or until PD or unacceptable toxicity or drug related DLT's for evaluation of pharmacokinetics (PK).
Period: Overall Study
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Started | 6 | 6 | 5 | 5
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 5 | 5
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Evidence of progressive disease | 4 | 6 | 4 | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all participants who received at least one dose of study drug.
Groups:
- Part A1: Eribulin Mesylate 1.1 mg/m^2: Participants received eribulin mesylate 1.1 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 4 cycles, or until PD or unacceptable toxicity or DLT's.
- Part A1: Eribulin Mesylate PK Expansion: Participants received eribulin mesylate 1.4 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 2 cycles, or until PD or unacceptable toxicity or drug related DLT's for evaluation of PK.
- Total: Total of all reporting groups
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion | Total
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (3.52) | 10.7 (2.25) | 13.0 (3.24) | 12.6 (5.50) | 12.5 (3.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 2 | 10
  Male | 5 | 2 | 2 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 6 | 4 | 4 | 4 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 5 | 5 | 4 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Eribulin Mesylate
Description: MTD: maximum dose at which <one third participants had DLT in Cycle 1. DLT: Grade 3/4 drug-related non hematological toxicity (except Grade 3 nausea, vomiting of <3 days, Grade 3 liver enzyme elevation with alanine transaminase/aspartate transaminase and gamma glutamyl transferase that returned to Grade <=1 or baseline prior to next dose; Grade 3 fever, infection, hypophosphatemia, hypokalemia, hypocalcemia/hypomagnesemia responsive to oral supplementation). Non-hematological toxicity causing >=14 days delay between treatment cycles. Haematological DLTs included: Grade 4 neutropenia/platelets<75,000/mm^3 on Day 8 that does not resolve to absolute neutrophil count >=750/mm^3 and platelets>=75,000/mm^3 by Day 11, neutropenia for >7 days; platelet count <25,000/mm^3, or required platelet transfusion, on 2 separate days within 7-day period;Grade 3 thrombocytopenia complicated by bleeding and/or required platelet transfusion;myelosuppression causing >14 days delay between treatment cycles.
Time Frame: First dose of study drug (Baseline) up to Cycle 1 Day 21
Population: The dose evaluable set (DES) included all participants who were judged as DLT evaluable as recorded in the database. In order to be DLT evaluable, all participants had to complete Cycle 1.
Measure: Number; unit: mg/m^2
Groups:
- Part A1: All Participants: All participants received eribulin mesylate 1.1 mg/m^2 or 1.4 mg/m^2 or 1.8 mg/m^2 or 1.4 mg/m^2 in PK expansion, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to a maximum of 8 cycles or until PD or unacceptable toxicity or drug related DLT's.
Arm/Group | Part A1: All Participants
Number analyzed (Participants) | 20
mg/m^2 | 1.4

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as those adverse events (AEs) that occurred (or worsened, if present at Baseline) after the first dose of study drug through 30 days after the last dose of study drug. An AE was defined as any untoward medical occurrence in a participants or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. A SAE was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect.
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (Cycle 8 Day 38)
Population: The SAS included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
Participants
  TEAEs | 6 | 6 | 5 | 5
  SAEs | 2 | 1 | 3 | 4

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Values
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (Cycle 8 Day 38)
Population: The SAS included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Vital Sign Values
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (Cycle 8 Day 38)
Population: The SAS included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (EKG)
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (Cycle 8 Day 38)
Population: The SAS included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
Participants
  >30 millisecond (msec) | 1 | 1 | 1 | 0
  >60 msec | 0 | 1 | 0 | 0

6. Primary Outcome: T1/2: Terminal Half-life for Eribulin Mesylate
Time Frame: Day 1 predose and at 10, 30 minutes, 1, 2, 4, 6, 24, 48, 72, 96 or 120 hours post-dose
Population: The pharmacokinetic analysis set (PAS) included all participants who had sufficient PK data to derive at least one PK parameter. The PAS where data at specified timepoints was available.
Measure: Median (Full Range); unit: hours
Groups:
- Part A1: Eribulin Mesylate 1.1 mg/m^2: Participants received eribulin mesylate 1.1 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up 4 cycles, or until PD or unacceptable toxicity or DLT's.
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 3 | 6 | 5 | 4
hours | 37.00 [29.6 to 38.9] | 38.60 [23.3 to 44.3] | 44.00 [30.6 to 56.5] | 33.25 [30.2 to 45.9]

7. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Eribulin Mesylate
Time Frame: Day 1 predose and at 10, 30 minutes, 1, 2, 4, 6, 24, 48, 72, 96 or 120 hours post-dose
Population: The PAS included all participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
nanogram/milliliter (ng/mL) | 353.8 (59.24) | 472.3 (158.23) | 382.6 (296.97) | 382.8 (247.05)

8. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Eribulin Mesylate
Time Frame: Day 1 predose and at 10, 30 minutes, 1, 2, 4, 6, 24, 48, 72, 96 or 120 hours post-dose
Population: The PAS included all participants who had sufficient PK data to derive at least one PK parameter.
Measure: Median (Full Range); unit: hours
Groups:
- Part A1: Eribulin Mesylate 1.1 mg/m2: Participants received eribulin mesylate 1.1 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 4 cycles, or until PD or unacceptable toxicity or DLT's.
- Part A1: Eribulin Mesylate 1.4 mg/m2: Participants received eribulin mesylate 1.4 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 8 cycles, or until PD or unacceptable toxicity or drug related DLT's.
- Part A1: Eribulin Mesylate 1.8 mg/m2: Participants received eribulin mesylate 1.8 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 5 cycles, or until PD or unacceptable toxicity or drug related DLT's.
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m2 | Part A1: Eribulin Mesylate 1.4 mg/m2 | Part A1: Eribulin Mesylate 1.8 mg/m2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
hours | 0.170 [0.12 to 0.32] | 0.170 [0.12 to 0.22] | 0.370 [0.08 to 0.50] | 0.300 [0.17 to 0.32]

9. Primary Outcome: AUC 0-t: Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for Eribulin Mesylate
Time Frame: Day 1 predose and at 10, 30 minutes, 1, 2, 4, 6, 24, 48, 72, 96 or 120 hours post-dose
Population: The PAS included all participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: hour * nanogram per milliliter (h*ng/mL)
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
hour * nanogram per milliliter (h*ng/mL) | 744.0 (353.03) | 758.2 (303.38) | 1363.0 (1378.53) | 1010.8 (538.94)

10. Primary Outcome: AUC 0-inf: Area Under the Concentration-time Curve From Zero (Pre-dose) Extrapolated to Infinite Time for Eribulin Mesylate
Time Frame: Day 1 predose and at 10, 30 minutes, 1, 2, 4, 6, 24, 48, 72, 96 or 120 hours post-dose
Population: The PAS included all participants who had sufficient PK data to derive at least one PK parameter. The PAS where data at specified timepoints was available.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 3 | 6 | 5 | 4
h*ng/mL | 654.3 (342.72) | 830.5 (331.14) | 1556.6 (1619.37) | 907.8 (493.59)

11. Primary Outcome: CL: Clearance for Eribulin Mesylate
Time Frame: Day 1 predose and at 10, 30 minutes, 1, 2, 4, 6, 24, 48, 72, 96 or 120 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: milliliter per hour (mL/h)
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 3 | 6 | 5 | 4
milliliter per hour (mL/h) | 2226.7 (957.10) | 1951.7 (469.27) | 2483.8 (1190.94) | 2348.8 (1437.56)

12. Primary Outcome: Vd: Volume of Distribution for Eribulin Mesylate
Time Frame: Day 1 predose and at 10, 30 minutes, 1, 2, 4, 6, 24, 48, 72, 96 or 120 hours post-dose
Population: The PAS included all participants who had sufficient PK data to derive at least one PK parameter. The PAS where data at pacified timepoints was available.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 3 | 6 | 5 | 4
milliliter | 75966.7 (34322.34) | 66766.7 (32230.40) | 89840.0 (43363.96) | 77525.0 (39176.64)

13. Secondary Outcome: Number of Participants With Best Overall Response
Description: Best Overall Response (BOR): best response recorded from start of study treatment until disease progression (PD) or recurrence based on response evaluation criteria in solid tumors (RECIST) version 1.1 for target and non-target lesions. Participants with evaluable disease were also eligible for assessment.
Time Frame: First dose of study drug (Baseline) up to approximately Cycle 8 (21-days treatment cycle)
Population: The SAS included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m2 | Part A1: Eribulin Mesylate PK Expansion
Number analyzed (Participants) | 6 | 6 | 5 | 5
Participants
  Stable Disease | 1 | 1 | 1 | 0
  Partial Response | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (Cycle 8 Day 38)
Groups:
- Part A1: Eribulin Mesylate 1.1 mg/m^2: Participants received eribulin mesylate 1.1 milligram mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 4 cycles, or until PD or unacceptable toxicity or DLT's.
- Part A1: Eribulin Mesylate PK Expansion: Participants received eribulin mesylate 1.8 mg/m^2, intravenously over 2 to 5 minutes on Days 1 and 8 of each 21-day treatment cycle for up to 2 cycles, or until PD or unacceptable toxicity or drug related DLT's for evaluation of PK.
Arm/Group | Part A1: Eribulin Mesylate 1.1 mg/m^2 | Part A1: Eribulin Mesylate 1.4 mg/m^2 | Part A1: Eribulin Mesylate 1.8 mg/m^2 | Part A1: Eribulin Mesylate PK Expansion
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 3/5 | 4/5
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A1: Eribulin Mesylate 1.1 mg/m^2 (N=6) | Part A1: Eribulin Mesylate 1.4 mg/m^2 (N=6) | Part A1: Eribulin Mesylate 1.8 mg/m^2 (N=5) | Part A1: Eribulin Mesylate PK Expansion (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A1: Eribulin Mesylate 1.1 mg/m^2 (N=6) | Part A1: Eribulin Mesylate 1.4 mg/m^2 (N=6) | Part A1: Eribulin Mesylate 1.8 mg/m^2 (N=5) | Part A1: Eribulin Mesylate PK Expansion (N=5)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 4 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2 | 2
Fatigue (General disorders) | 2 | 1 | 2 | 2
Malaise (General disorders) | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 4 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 2 | 1
Blood albumin decreased (Investigations) | 2 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 1 | 1
Blood chloride decreased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 2 | 1
Blood sodium decreased (Investigations) | 3 | 2 | 0 | 1
Blood urine present (Investigations) | 0 | 1 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 1 | 2
Haemoglobin decreased (Investigations) | 3 | 3 | 4 | 0
Lymphocyte count decreased (Investigations) | 4 | 3 | 3 | 4
Neutrophil count decreased (Investigations) | 5 | 2 | 4 | 2
Platelet count decreased (Investigations) | 1 | 2 | 4 | 2
Protein urine present (Investigations) | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 2 | 0
White blood cell count decreased (Investigations) | 5 | 5 | 5 | 4
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
In Part A2, the study was open for the enrolment of infant participants of less than 12 months of age, however no participants were enrolled into this part.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No